

# RÉSUMÉ DU PROTOCOLE POUR LES RECHERCHES MENTIONNÉES AU 30 DE L'ARTICLE L. 1121-1 DU CODE DE LA SANTÉ PUBLIQUE NE COMPORTANT QUE DES QUESTIONNAIRES OU DES ENTRETIENS

| Titre de la recherche | | Evaluation de la connaissance de son statut vaccinal et du rapport à la vaccination chez les patients à l'hôpital de Melun |
|---|---|---|
| Titre abrégé de la recherche | | Statuvax pat |
| Numéro d'enregistrement (ID-RCB) | | 2023-A01028-37 |
| Date et numéro de version du Résumé: | | Version 4 du 16/09/2023 |
| Date et numéro de version de la note d'information (joindre ce document) : | | Version 4 du 16/09/2023 |
| Date et numéro de la version des questionnaires et/<br>ou de la trame des entretiens (à joindre ces<br>documents) : | | Version 6 du 16/09/2023 |
| Conformité de cette demande d'avis avec la procédure prévue au <u>II de l'article R. 1123-20 du code de la santé publique</u> (une réponse négative à l'un des quatre critères ci-dessous signifie que vous ne relevez pas de cette procédure) : | | |
| Cette recher | che comporte uniquement des données recue | illies par questionnaire (s) ou entretien (s): |
| | ⊠ OUI | |
| Cette recherche n'a aucune conséquence pour les personnes participantes que ce soit en termes de sécurité ou de modification de la prise en charge habituelle : | | |
| Cette recherche est dénuée de risque et les inconvénients pour les personnes participantes à la recherche sont négligeables : | | |
| | OUI<br>NON | |
| Le recueil et le traitement des données mis en œuvre dans cette recherche sont conformes à la méthodologie de référence MR003 homologuée par la CNIL : | | |
| $\boxtimes$ | OUI | |
| | NON | |





| Informations administratives | |
|---|---|
| Promoteur: | Groupe Hospitalier Sud Ile de France |
| Courriel : | drc.promotion@ghsif.fr |
| Adresse : | 270 avenue Marc Jacquet 77000 Melun |
| Téléphone : | 01 81 74 17 17 |
| Responsable Unité de Recherche Clinique | M. Arezki AGHER |
| Courriel | arezki.agher@ghsif.fr |
| Téléphone/Fax | Tel: 01 81 74 22 28 Fax: 01 81 74 25 59 |
| Investigateur ou, le cas échéant, investigateur coordonnateur | |
| Nom, Prénom et Fonction : | Dr Coralie Noel, Praticien Hospitalier en Hygiène<br>Hospitalière au Centre Hospitalier de Melun |
| Courriel : | coralie.noel@ghsif.fr |
| Adresse du lieu principal de la recherche : | 270 avenue Marc Jacquet 77000 Melun |
| Téléphone : | 01 81 74 21 27 |
| Nombre de centre si recherche<br>multicentrique : | 1 centre |

### Contexte et justification de la recherche

Le contexte de la recherche

Les couvertures vaccinales des personnes adultes en France sont médiocres : seulement 44% des personnes âgées de 65 ans et plus sont à jour vis-à-vis de la vaccination diphtérie, tétanos et poliomyélite infectieuse (1), et dans une étude plus ancienne en 2002, chez les personnes âgées de 16 ans et plus, de 71,2% contre le tétanos, 41.9% contre la poliomyélite infectieuse et 33.7% contre la diphtérie (2). D'autres vaccinations peuvent être recommandées selon les comorbidités des personnes, tel que la vaccination antipneumococcique, et la couverture vaccinale est parfois très basse selon les pathologies (contre le pneumocoque, moins de 2% des diabétiques sont correctement immunisés) (3), alors que les couvertures vaccinales contre le SARS-CoV-2 sont bien meilleures (plus de 90% chez les diabétiques par exemple) selon les données de l'Assurance maladie (4), sous



l'influence d'une politique vaccinale proactive, voire coercitive.

L'hospitalisation est rarement le moment où les patients peuvent bénéficier d'une évaluation de leur statut vaccinal, et ce rôle est bien souvent laissé au médecin traitant, dont les missions de prévention sont souvent reléguées au second plan en raison d'une pénurie globale, et particulièrement marquée sur le territoire du Sud Seine-et-Marne.

Dans le cadre de la manifestation nationale « Semaine Européenne de la Vaccination » portée par le Ministère de la Santé et de la Prévention, nous proposons un questionnaire à un échantillon de patients hospitalisés dans notre hôpital sur la connaissance de leur statut vaccinal et évaluer leur rapport à la vaccination.

- 1. Institut National de Veille Sanitaire (InVS). Enquête nationale de couverture vaccinale, France, janvier 2011. Couverture vaccinale contre la grippe saisonnière dans les groupes cibles et mesure de l'efficacité vaccinale. Couverture vaccinale par les vaccins diphtérie-tétanos-poliomyélite (dTP) et... [Internet]. 2011 [cité 11 avr 2023] p. 21. Disponible sur : https://www.santepubliquefrance.fr/content/download/1817 15/2304769?version=1
- 2. Guthmann JP, Fonteneau L, Antona D, Lévy-Bruhl D. La couverture vaccinale diphtérie, tétanos, poliomyélite chez l'adulte en France : résultats de l'enquête Santé et Protection Sociale, 2002. Bull Epidemiol Hebd. déc 2007;(51-52):441-5.
- 3. Wyplosz B, Fernandes J, Sultan A, Roche N, Roubille F, Loubet P, et al. Pneumococcal and influenza vaccination coverage among at-risk adults: A 5-year French national observational study. Vaccine. 5 août 2022; 40(33):4911-21.
- 4. Data Vaccin Covid (Assurance Maladie) [Internet]. [cité 11 avr 2023]. Disponible sur: https://datavaccincovid.ameli.fr/pages/home/

Les hypothèses de la recherche

35% des patients pensent connaître leur statut vaccinal.

### Objectifs et critères de jugement

Objectif principal de la recherche et critère de jugement principal

Evaluation du taux de connaissance de son propre statut vaccinal chez les patients hospitalisés au CH de Melun.



## Objectif (s) secondaire (s) et critère (s) de jugement secondaires éventuels

Evaluation du rapport qu'ont les patients hospitalisés vis-à-vis de la vaccination en général. Evaluer par le nombre de patients qui souhaitent se mettre à jour de leur vaccination.

Observer l'influence des différents facteurs (sexe, métier, présence ou non de médecin traitant, Etat de mal chronique) sur le statut vaccinal à Melun.

### Organisation de l'étude

A. Description synthétique du schéma d'étude

☐ si non validé, justifier :

Questionnaire administré au patient au cours de son hospitalisation. Patients aléatoirement à l'aide du DIM de l'hôpital au début de la semaine de l'enquête.

Patients qui seront aléatoirement choisi dans chacun des 10 services de soins du CH de Melun ((Médecine interne, maladies infectieuses, gastro entérologie, pneumologie, chirurgie, médecine BCR, cardiologie, néphrologie, soins de suite et réadaptation et gériatrie) et accompagnés pour remplir un questionnaire mis en place par USP et EOH du CH de Melun.

| | gériatrie) et accompagnés pour remplir un questionnaire mis en place par USP et EOH du CH de Melun. |
|---|---|
| B. Méthodologie des questionnaires/ entretiens | |
| - <b>Questionnaire (s)</b> Oui | |
| Modalités de passation : | |
| Questionnaire administré par : | |
| ☐ courrier | |
| □ internet | |
| ☐ téléphone | |
| <ul><li>autre (préciser)</li></ul> | |
| Questionnaire administré en : | |
| □ une fois | |
| <ul> <li>plusieurs fois (préciser le nombre de passa</li> </ul> | ition) : |
| Type de questionnaires : | |
| ☒ si validé, indiquer l'origine de la validation | : USP et EOH |



| C. | Trame de l'analyse statistique et/ ou références du |
|----|-----------------------------------------------------|
| | biostatisticien responsable : |

Statistiques descriptives (fréquences, moyennes, écartstypes). Analyse des variables indépendantes par le test de Chi-2.

| Informations relatives à la mise en œuvre de la recherche | |
|---|---|
| A. Type de lieu où doit se dérouler la recherche | Service hospitalier |
| B. Durée prévisionnelle de la recherche : | 1 mois |
| C. Durée prévisionnelle de participation par personne : | 20 minutes |
| D. La recherche implique-t-elle en plus un recueil de données rétrospectives : | □ OUI<br>⊠ NON |
| E. Personnes incluses dans la recherche | |
| Nombre de personnes interrogées : | 140 patients |
| Critères d'inclusion : | Patient adulte (Age ≥ 18 ans) , lieu de résidence principale<br>en France, hospitalisé dans un service du CH de Melun,<br>pouvant parler et comprendre le français et non dément |
| Critères de non-inclusion : | Ne parle pas français ou démence<br>Refus du patient de participer à l'étude. |
| Critères d'exclusion secondaire : | Moins de 18 ans |
| La recherche inclut-elle des personnes ne présentant aucune affection ? | non |
| Modalités de recrutement des personnes interrogées : | Tirage au sort de 14 patients dans services de soins et questionnaire réalisé si répond aux critères inclusion |
| Modalités d'information et de traçabilité de la non-<br>opposition : | Formulaire signé d'opposition |







| F. Inconvénients pour les personnes incluses dans la recherche | |
|---|---|
| Durée prévisionnelle du recueil de données par entretien ou questionnaire pour un participant : | 20 min |
| Durée prévisionnelle totale de participation à la recherche pour un participant si le recueil de données est réalisé en plusieurs fois (durée entre l'inclusion et le dernier recueil de données) : | 20 min |
| Temps de transport maximal estimé pour les participants si applicable : | N/A |